CLINICAL TRIAL: NCT07028307
Title: Effects of Kinesio Taping and Breathing Exercises in Individuals With Hyperkyphosis
Brief Title: Effect of Kinesio Tape and Breathing Exercises in Hyperkyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYPHSZ-2025
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Breathing Exercise; Pranayama; Kinesio Taping; Hyperkyphosis
Keywords: kinesiotaping; pranayama; hyperkyphosis; breathing exercise
MeSH Terms: conditions — Kyphosis | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises Group (Active Comparator): The breathing exercises applied included yogic pranayama techniques and were performed face to face one day a week and followed with an exercise diary to indicate that they continued these exercises on the remaining days of the week, for a total of 5 days a week and 4 weeks. Reminder messages for the exercises were sent through the WhatsApp group opened with all participants included in the study. In the first session, patient education was given about diaphragmatic breathing and its importance. The breathing techniques applied included Ujjai, Sukha Pranayama and Nadi Shodhana techniques.
  Interventions: Other: Breathing Exercises
- Breathing Exercises + Kinesio Taping Group (Active Comparator): In addition to the breathing techniques and patient education applied in the breathing exercises group; kinesiotape application for hyperkyphosis was applied by the same physiotherapist once a week for 4 weeks.
  Interventions: Other: Breathing Exercises + Kinesio Taping Group

INTERVENTIONS:
Other: Breathing Exercises — Ujjai: While the mouth is closed, a hissing sound is made until the space between the throat and lungs is filled with breath, and a slow and deep inhalation is made. Then, without holding the breath, a long and full exhalation is made through a partially closed glottis and a slight laryngeal muscle contraction, and the same sound is made. In each session, two sets of ujjayi technique were applied, with an inhalation:exhalation ratio of 1:2 and 10 respiratory cycles, with a 1-minute rest period between sets.
  Sukha Pranayama: Applied for 5 minutes with a 5:5 inhalation:exhalation ratio of 6 breaths per minute.
  Nadi Shodhana: After closing the right nostril with the thumb of the right hand, a slow and deep inhalation is performed through the left nostril. After maximum inhalation, without holding the breath, the left nostril is closed with the fourth finger of the right hand and a full exhalation is performed through the right nostril. Maintaining the closed position of the left nostr
  Arms: Breathing Exercises Group
Other: Breathing Exercises + Kinesio Taping Group — The tape was not removed for 5 days from the day of the procedure, but was removed after the 5th day, allowing the skin to rest for 2 days, and then repeated for 4 weeks with a new kinesio tape application. The tapes of those who stated that there was wear or tear on the tape were renewed within a week. After the skin was cleaned with alcohol, the kinesio tape application was applied bilaterally as an I tape with 25-50% tension on the paraspinal muscles from the 7th cervical vertebra to the 12th thoracic vertebra. The I tape was applied horizontally with 50% tension to the point where the kyphotic area was clearly observed. All strips were rubbed to increase adhesion to the skin and activate the tape.
  Arms: Breathing Exercises + Kinesio Taping Group

SUMMARY:
The aim of this study was to evaluate the effects of breathing exercises alone and in combination with kinesiotape application on pain experience, postural alignment, sleep quality, anxiety level, and respiratory capacity in university students with thoracic hyperkyphosis. A total of 30 university students aged between 19-30 with complaints of back pain and increased kyphosis were included in the study and the participants were divided into 2 groups. Breathing exercises included yogic pranayama techniques and were performed 5 days a week for 4 weeks. In the breathing exercises and kinesiotape group, in addition to the breathing exercises applied; kinesiotape application for hyperkyphosis was applied once a week for 4 weeks. Within the scope of the study, participants' posture, respiratory capacity, pain level, anxiety level and functional posture parameters were evaluated.

DETAILED DESCRIPTION:
Today, back pain has become one of the most common health problems encountered by physiotherapists. In the emergence of back pain; structural, functional and mechanical disorders of the spine, biological factors such as obesity, psychological disorders such as anxiety and depression, and social factors such as age, gender, economic status and working conditions play an important role. In addition, staying inactive for long hours, incorrect sitting positions, lifting heavy loads or repetitive incorrect movements can also cause back pain to worsen. Today's living conditions, with the decrease in physical activity and increase in stress, cause back pain to become more common. In order to prevent this situation, it is very important to do regular exercise, gain posture habits suitable for body mechanics and create ergonomic working conditions. One of the most important causes of back pain is posture disorder. Bad posture disrupts the equal distribution of compressive and tension forces that should be balanced on the body axis, causing various structural problems in the spine. As a result, nerve roots can be compressed, intervertebral foramina can narrow, and repetitive tensions can occur in the muscles, causing back pain. Bad posture, which is considered inadequate body posture, causes muscles, bones, and other structures to work excessively, paving the way for serious problems to develop in the body over time. Smartphone addiction in university students can lead to many physical ailments such as back, waist, and neck pain. It has been observed that back pain in university students is associated with anxiety and depressive symptoms. However, back pain caused by kyphosis can also affect psychological status. Schmidt stated that back pain is more severe in patients who are insecure and uncompliant, and that these patients are individuals who are subjectively prone to burnout. Occiput-wall distance (OWD), which is a measure of kyphosis, has been associated with posture disorder, osteoporosis, disability and depression. Techniques such as kinesio tape, postural exercises, manual therapy, Schroth method and stretching exercises can be applied in the treatment of kyphosis. It has been explained that the application of kinesio tape in university students has positive effects in reducing the thoracic kyphosis angle and increasing postural awareness.Breathing exercises are an effective method for correcting posture and improving spinal health in individuals with increased kyphosis. Kyphosis usually results in posture disorders as a result of excessive curvature in the upper part of the spine. Breathing exercises encourage the correct use of the diaphragm in particular and help correct body posture. Deep breathing and activating the diaphragm muscles make it easier to keep the spine upright, strengthen the back muscles and make the body more stable. Today, we are encountering an increase in posture disorders more commonly every year, especially among university students with a young population. It is very important to determine the level of postural problems and pain experience that develop and are likely to progress in university students and the approaches to prevent them. When the literature is examined, there is no study showing the effects of the combined application of kinesiotape and breathing exercises to individuals with postural kyphosis. In this context, the aim of the study is to evaluate the effects of the use of breathing exercises alone and the combined use of breathing exercises and kinesiotape application on pain experience, postural improvement, sleep quality, anxiety level and respiratory capacity in university students with thoracic hyperkyphosis.

ELIGIBILITY:
Inclusion Criteria:

* University students
* Those with hyperkyphosis
* Those who volunteer to participate in the study

Exclusion Criteria:

* Respiratory diseases: Individuals diagnosed with asthma, COPD, interstitial lung diseases and other chronic respiratory diseases
* Smoking
* Surgical history
* Pharmacological treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
The New York Posture Rating | Baseline and week 4
  It is an assessment tool developed to determine the posture disorders of individuals. It was first published in 1958 and allows the body to be analyzed from anterior (front) and lateral (side) perspectives by dividing it into 13 different regions.
The McGill Pain Questionnaire | Baseline and week 4
  The questionnaire consists of four main sections. At the beginning of the form, there is information about the patient's medical diagnosis and current problem, the analgesic drugs used and their type and dosage, as well as the patient's perception of pain, the location of the pain, its characteristics, its relationship with time and its severity.
Pittsburgh Sleep Quality Index | Baseline and 4 week
  The scale consists of 24 questions in total. The scale consists of 7 components that evaluate sleep quality: subjective sleep quality, sleep latency (time to fall asleep), sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. A high total score from the scale indicates poor sleep quality. A score of 5 or more on the Pittsburgh Sleep Quality Scale indicates poor sleep quality.
Beck Anxiety Inventory | Baseline and week 4
  It was developed by Beck et al. (1988) to measure anxiety severity and consists of 21 items. The total score of the scale varies between 0 and 63.
Body Oxygen Level Test | Baseline and week 4
  The BOLT test is usually related to the breathing pattern, breath holding time and oxygen level. A low BOLT score of 10-20 seconds indicates poor respiratory capacity and inadequate oxygen intake, while 25-40 seconds is normal, and 40 and above indicates a high BOLT score, which means improved oxygen capacity.
C7- Wall Distance | Baseline and week 4
  It is a valid and reliable testing method that measures the perpendicular distance from the C7 spinous process to the wall.
Occiput Wall Distance:OWD | Baseline and week 4
  Participants are asked to touch their occiput to the wall while their backs and heels are against the wall and their heads are looking forward. The distance is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Health and Technology University, Istanbul, Beyoğlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No